CLINICAL TRIAL: NCT05737043
Title: Comparison of the Modified Myocardial Performance Index and Epicardial Thickness in Cases With Idiopathic Polyhydramnios and in Healthy Normal Pregnancies
Brief Title: Modified Myocardial Performance Index and Epicardial Thickness in Cases With Idiopathic Polyhydramnios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, şükran doğru, md, Necmettin Erbakan University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2023/4145(10675: neu)
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Fetal Diagnose; Fetal Cardiac Disorder
Keywords: polyhidramnios, epicard, myocardial performance index

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myocardial performance and epicard thickness in case with polyhidramnios (Placebo Comparator): we will do a fetal echo, and fetal screening with ultrasonography
  Interventions: Diagnostic Test: prenatal diagnose
- pregnant women with polyhidramios (Active Comparator)
  Interventions: Diagnostic Test: prenatal diagnose

INTERVENTIONS:
Diagnostic Test: prenatal diagnose — we will do a fetal echo in pregnant women with polyhidramnios

SUMMARY:
In cases diagnosed as idiopathic polyhydramnios and healthy pregnancy between 24-40 weeks (total number of cases (100-120)), prospective fetal echocardiography will be performed to evaluate MPI and EFT.

DETAILED DESCRIPTION:
: gestational week, maternal age, amniotic fluid index measurement, modified myocardial performance in fetal echo and epicardial thickness of all cases will be evaluated. week of pregnancy, body mass index, fetal biometry, umbilical artery doppler, middle cerebral artery doppler measurements will be taken. Birth weight and fetal intensive care hospitalizations at the birth week of all cases will be recorded. All data will be evaluated with the appropriate statistical method.

ELIGIBILITY:
Inclusion Criteria: 24-40 weeks gestational age, polyhydramnios and healthy pregnancy -

Exclusion Criteria: multıpl pregnancy, fetal anomaly, growth restriction, maternal chronic disease

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
neonatal and fetal outcome | 1 year
  Do epicardial thickness and myocardial performance index determine fetal outcome in cases with polyhdramnios?

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I want to share it as an article when the results are collected